CLINICAL TRIAL: NCT05959343
Title: A Prospective, Randomized Controlled Trial Comparing the Outcomes of an Enhanced Recovery After Surgery (ERAS) Program With Non-ERAS Care in Patients Undergoing Oblique Lumbar Interbody Fusion (OLIF)
Brief Title: Enhanced Recovery After Surgery in Oblique Lumbar Interbody Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Medical Research Collaborating Center, Seoul, Korea (Other); Armed Forces Capital Hospital, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Chi Heon Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-2305-085-1423
Record Dates: First submitted 2023-06-22; First posted 2023-07-25 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Enhanced Recovery After Surgery; Spinal Fusion; Lumbar Spinal Stenosis; Lumbar Spondylolisthesis
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): The experimental group will be implemented with the ERAS Clinical Pathway (ERAS CP)
  Interventions: Behavioral: Enhanced Recovery After Surgery program for Oblique Lumbar Interbody Fusion
- Control group (No Intervention): The control group will not be implemented with the ERAS CP

INTERVENTIONS:
Behavioral: Enhanced Recovery After Surgery program for Oblique Lumbar Interbody Fusion — In the ERAS CP group, the components of the ERAS are protocolized and implemented as a clinical pathway
  Arms: ERAS group

SUMMARY:
This study is a randomized controlled non-inferiority trial designed to evaluate the impact of implementing the 'Early Recovery After Surgery Clinical Pathway (ERAS CP)' on patient-reported pain levels at the time of discharge following Oblique Lumbar Interbody Fusion (OLIF) surgery

DETAILED DESCRIPTION:
Currently, the effectiveness of the ERAS has been widely confirmed in patients undergoing colorectal resection, and it has been verified to reduce length of hospital stay and complications. However, the ERAS protocol for lumbar fusion surgery is based on a few retrospective studies and remains a consensus statement. Recent retrospective studies targeting patients undergoing lumbar fusion surgery reported that implementing ERAS could accelerate post-operative functional recovery and reduce hospital stay. However, there is still a lack of high-quality evidence based on prospective studies.

Lumbar fusion surgery is known for potentially leading to severe postoperative pain, which poses challenges in consistently applying ERAS components, such as early ambulation or active oral feeding, after surgery. In light of this, the present study aims to validate the non-inferiority of pain levels at discharge within the ERAS group and to reconfirm the effects of ERAS as observed in retrospective studies.

Patients admitted for OLIF will be consecutively screened for eligibility. A computer-generated block randomization will be executed at a 1:1 ratio. In the ERAS group, patients will receive comprehensive education about the treatment process, and a clinical pathway that includes active ambulation and pain control will be protocolized and implemented. Should non-inferiority be demonstrated in both intent-to-treat and per-protocol analyses, non-inferiority will be declared.

ELIGIBILITY:
Inclusion Criteria:

1. Lumbar degenerative disease, requiring interbody fusion of 1-2 segments between L2 and S1
2. Capability of independent (or assisted) ambulation for at least 30 minutes with

   1. Taking intermittent breaks
   2. Enduring any discomfort
3. Voluntary informed consent to participate in the study.

Exclusion Criteria:

1. Previous history of lumbar interbody fusion
2. Manual Muscle Testing grade 3 or below
3. Neuropsychiatric disorders such as major depressive disorder
4. Musculoskeletal disorders other than lumbar degenerative diseases (inflammatory, myopathic, infections, etc.)
5. Diagnosis of malignant neoplasm
6. Refusal to participate in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale for back pain and leg pain | 1 day at discharge
  Pain intensity will be recorded on a scale from 0 to 10, with 0 indicating no pain and 10 indicating the maximum pain imaginable.

SECONDARY OUTCOMES:
First ambulation time | about postoperative 0~1 day (ex. 4 hours after surgery, 18 hours after surgery)
  The time at which a patient first began ambulation after returning to the ward from the operating room
First self-urination time | about postoperative 0~1 day (ex. 4 hours after surgery, 18 hours after surgery)
  The time at which self-voiding was first initiated after the removal of foley catheter
Numeric Rating Scale for back pain and leg pain during inhospital status | Daily measurement through the hospitalization period for surgery(ex. at postoperative 1day, at postoperative 2day), Postoperative 1-month
  Pain intensity will be recorded on a scale from 0 to 10, with 0 indicating no pain and 10 indicating the maximum pain imaginable.
Total analgesic consumption | Daily measurement through the hospitalization period for surgery(ex. at postoperative 1 day, at postoperative 3 day)
  Total dose analgesic used during inhospital status
Patient satisfaction scale | 1 day at discharge, Postoperative 1-month
  We survey patients using a 4-point scale to gauge their overall satisfaction with the treatment process. On this scale, 4 represents 'very satisfied,' 3 is 'satisfied,' 2 is 'dissatisfied,' and 1 indicates 'very dissatisfied.
Rate of complication related to surgery | through study completion, an average of 6 month
  We investigate complications related to the surgery. Such complications include vascular damage, ureteral injury, abdominal wall injury, herniation, sympathetic nerve chain damage, leg weakness, and surgical wound infections.
Rate of medical complication | through study completion, an average of 6 month
  We examine postoperative internal medicine complications. These complications encompass cardiovascular issues, gastrointestinal disturbances, non-surgical site infections, renal problems, and electrolyte abnormalities.
30-day readmission | upto postoperative 30 days
  Any 30-day readmission after surgery
medial cost | postoperative 1-month
  The total medical cost incurred during the in-hospital stay for the surgery will be calculated
length of hospital stay | postoperative 1-month
  length of the hospitalization days

CONTACTS AND LOCATIONS:
Overall Officials: Chi Heon Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after primary analysis
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After analysis
Access Criteria: With any reasonable requeset

REFERENCES:
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Debono B, Wainwright TW, Wang MY, Sigmundsson FG, Yang MMH, Smid-Nanninga H, Bonnal A, Le Huec JC, Fawcett WJ, Ljungqvist O, Lonjon G, de Boer HD. Consensus statement for perioperative care in lumbar spinal fusion: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Spine J. 2021 May;21(5):729-752. doi: 10.1016/j.spinee.2021.01.001. Epub 2021 Jan 12. PMID 33444664
- [Result] Porche K, Yan S, Mohamed B, Garvan C, Samra R, Melnick K, Vaziri S, Seubert C, Decker M, Polifka A, Hoh DJ. Enhanced recovery after surgery (ERAS) improves return of physiological function in frail patients undergoing one- to two-level TLIFs: an observational retrospective cohort study. Spine J. 2022 Sep;22(9):1513-1522. doi: 10.1016/j.spinee.2022.04.007. Epub 2022 Apr 18. PMID 35447326
- [Result] Porche K, Samra R, Melnick K, Brennan M, Vaziri S, Seubert C, Polifka A, Hoh DJ, Mohamed B. Enhanced recovery after surgery (ERAS) for open transforaminal lumbar interbody fusion: a retrospective propensity-matched cohort study. Spine J. 2022 Mar;22(3):399-410. doi: 10.1016/j.spinee.2021.10.007. Epub 2021 Oct 21. PMID 34687905